CLINICAL TRIAL: NCT02307708
Title: Reeducation of Chronic Achilles Tendinopathy by Wearing Shoes Inclined Versus Reeducation by Kinesitherapy
Acronym: TARCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties (few patients meeting inclusion criteria, refusal of patients to stop sport activities during 6 weeks,...)
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC13_0043
Record Dates: First submitted 2014-07-25; First posted 2014-12-04 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Tendinopathy; Rupture of Achilles Tendon; Chronic Disease
MeSH Terms: conditions — Tendinopathy; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8° incline shoe (Experimental): The shoe is inclined from front to back and from top to bottom of 8 °. This causes a controlled and an eccentric contraction during the passage.
  During the walk we will have:
  In support tardigrade : an ankle dorsiflexion with a stretching the Achilles tendon (eccentric contractions).
  In support digitigrade: plantar flexion of ankle with a muscle contraction of triceps surae (concentric contraction).
  Interventions: Device: 8° incline shoe
- kinesitherapy (Active Comparator): The patient performs its home therapy and consults his physiotherapist once a week according to the protocol Stanish
  Interventions: Other: kinesitherapy

INTERVENTIONS:
Device: 8° incline shoe — Wearing inclined shoes for 6 weeks, walking 15 minutes (2 times/day).
  The shoe is inclined from front to back and from top to bottom of 8 °. This causes a controlled and an eccentric contraction during the passage.
  During the walk we will have:
  In support tardigrade : an ankle dorsiflexion with a stretching the Achilles tendon (eccentric contractions).
  In support digitigrade: plantar flexion of ankle with a muscle contraction of triceps surae (concentric contraction).
  Other Names: Wearing inclined shoes
  Arms: 8° incline shoe
Other: kinesitherapy — Daily eccentric contraction at home and once per week for 6 weeks with the physiotherapist
  Other Names: The kinesitherapy for the treatment of tendinopathy
  Arms: kinesitherapy

SUMMARY:
The purpose of the study is to compare the treatment by wearing shoes inclined at kinesitherapy because it is the first treatment offered by primary care physicians in chronic Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Disease: chronic Achilles tendinopathy de novo or recurrent confirmed by ultrasound
* Patients having signed the informed consent for the study participation
* Patients covered by medical insurance
* Patients having no behavioral disorders

Exclusion Criteria:

* History of rupture of the Achilles tendon (= stage 4)
* Antibiotic treatment tendinotoxique (Quinolones, ...)
* Inability to walk more than 30 minutes per day.
* Haglund Syndrome
* Treatment of tendinopathy or being older than six months
* Minors
* Major trust

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evolution of the American Orthopaedic Foot and Ankle Score (AOFAS) | at Day 0 and 12 weeks

SECONDARY OUTCOMES:
Evolution of amplitude to the tibio-tarsal | at 12 weeks
Pain Scores on the Visual Analog Scale | at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Rousseau, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - CHU de Nantes, Nantes
  - Nouvelles cliniques Nantaises, Nantes